CLINICAL TRIAL: NCT04276012
Title: Effectiveness of a Cardiovascular Risk Intervention Program in Patients With Schizophrenia: PRISCA Study
Brief Title: Effectiveness of a Cardiovascular Risk Intervention Program in Patients With Schizophrenia (PRISCA)
Acronym: PRISCA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dr. Pere Roura-Poch (Other)
Responsible Party: Sponsor-Investigator, Dr. Pere Roura-Poch, Epidemiologist, Consorci Hospitalari de Vic
Organization: Consorci Hospitalari de Vic (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AC-274
Record Dates: First submitted 2020-02-17; First posted 2020-02-19 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Schizophrenia; Cardiovascular Risk Factor
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention group will participate in different intervention strategy depending on the individual needs (psychoeducational, recommendations of life style and diet, medication adherence and changes in pharmacological strategy)
  Interventions: Other: Multifactorial intervention
- Control group (No Intervention): Usual clinical care

INTERVENTIONS:
Other: Multifactorial intervention — Psychoeducational intervention, recommendations on life style and diet, medication adherence and changes in pharmacological strategy
  Arms: Intervention group

SUMMARY:
The main objective is to determine the effectiveness of a program which consists of multidisciplinary, intensive and individualized interventions, carried out by a group of health professionals (psychiatrist, psychologist, mental health nurse, primary care doctors, pharmacist), during six-month, to improve the global cardiovascular risk (CVR) in patients with schizophrenia. Secondarily, will be analyzed the effectiveness of this program on improving the control in four selected cardiovascular risk factors: hypertension, hypercholesterolemia, hyperglycaemia and smoking, after 6 months Methods: randomized study with parallel assignment in two groups: control and intervention group, six-month follow-up. The eligible patients will be 130 adult (≥18 years) outpatients with a current diagnosis of schizophrenia who follow-up by health mental network in Catalonia, who presents at least bad control in one of the four selected cardiovascular risk factors. The intervention group will receive a multidisciplinary and individualized approach (psychoeducational, recommendations of life style and diet, medication adherence and changes in pharmacological strategy, depending on the individual needs assessing after cardiovascular risk screening. The control group will follow the standard management according to the primary care professionals' team.

Main measurements: the global CVR at baseline and at six-month follow-up through Framingham tables calibrated for the Catalan population (Registre Gironí del Cor, REGICOR). Secondary measures: they will be determined, at baseline and at six-month follow-up, four cardiovascular risk factors as well: hypertension, hypercholesterolemia, hyperglycaemia and smoking, according with the latest recommendations of the Program of preventive activities and health promotion (PAPPS) of the Spanish Society of Family and Community Medicine. Other measures: anthropometric parameters. Functional Assessment Screening Tool (FAST) and quality of life (EQ-5D).

ELIGIBILITY:
Inclusion Criteria:

adults (≥18 years of age), outpatient, current diagnostic of schizophrenia, follow-up by mental health network in Catalonia, signed informed consent.

Exclusion Criteria:

other severe mental illnesses different from schizophrenia, patients with intellectual disabilities or clinical acute psychotic relapse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2020-01-20 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-02-28 (Estimated)

PRIMARY OUTCOMES:
Changes in global cardiovascular risk | At six months
  Framingham tables calibrated for the Catalan population (Registre Gironí del Cor, REGICOR). The CVR was stratified into the following groups:<5%, low; 5-9%, moderate; 10-14%, high; and ≥15, very high.

SECONDARY OUTCOMES:
Changes in systolic/diastolic blood pressure | At six months
  mmHg
Changes in glycated haemoglobin | At six months
  Percentage of
Changes in cholesterolemia level and other lipids in blood | At six months
  mg/dL
Stopping tobacco | At six months
  Yes/No

CONTACTS AND LOCATIONS:
Locations (1):
- Vic Hospital Consortium, Vic, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Riera-Molist N, Assens-Tauste M, Roura-Poch P, Guimera-Gallent M, Santos-Lopez JM, Serra-Millas M, Frau-Rossello N, Gallego-Pena E, Foguet-Boreu Q. A Cardiovascular Risk Optimization Program in People With Schizophrenia: A Pilot Randomized Controlled Clinical Trial. J Psychiatr Pract. 2023 Nov 1;29(6):456-468. doi: 10.1097/PRA.0000000000000743. PMID 37948170